CLINICAL TRIAL: NCT02056795
Title: A Single Application of Electroacupuncture Improves Balance Greater Than Placebo Control in Subjects With Chronic Functional Ankle Instability
Brief Title: Study of Effects of Electroacupuncture on Balance in Subjects With Chronic Functional Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canadian Memorial Chiropractic College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 122017
Record Dates: First submitted 2014-01-24; First posted 2014-02-06 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Ankle Sprain
MeSH Terms: conditions — Ankle Injuries | interventions — Needles; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electroacupuncture (Experimental): Subjects will do balance assessment in lab. In treatment room, practitioner will clean insertion area with alcohol swab, allow adequate time to dry, and insert 2 Asia-Med Special No 16 (0.30x30mm) needles: one at proximal insertion of fibularis longus anterior to fibular neck, in proximity to common fibular nerve (GB-34); one over sinus tarsi and lateral ligaments of ankle mortise (GB-40). Needles will be inserted approximately 1-2cm, connected for 10 min at 2Hz to electrical stimulation (ITO ES-130, 500 ohm test load, 1 to 500Hz). Needles will disposed of in sharps container. Area will be wiped with long handled cotton swab, pressure will be applied for 2 seconds. Subjects will be asked to slowly get up from table and return to lab for second balance assessment.
  Interventions: Device: Asia-Med Special No 16 (0.30x30mm) needles
- Control (Sham Comparator): As with experimental group, controls will do balance assessment pre- and post-intervention. Streitberger placebo needles (Asia-Med, 0.03 x 30 mm), blunted with a telescoping mechanism, will be used. Subjects will feel slight prick, and shaft will telescope into handle, creating illusion of skin penetration. Needles will be held in place by plastic ring covered by a bandage. They are validated for blinding. They will be placed over non-traditional acupuncture points on medial aspect of leg, in direct opposition to treatment group needles. Needle placement is not intended to produce therapeutic outcome. The needles will be connected to a wire, which will be turned on for 10 minutes but no stimulation will be felt.
  Interventions: Device: Streitberger placebo needles (Asia-Med, 0.03 x 30 mm)

INTERVENTIONS:
Device: Asia-Med Special No 16 (0.30x30mm) needles — Subjects will do balance assessment in lab. In treatment room, practitioner will clean insertion area with alcohol swab, allow adequate time to dry, and insert 2 Asia-Med Special No 16 (0.30x30mm) needles: one at proximal insertion of fibularis longus anterior to fibular neck, in proximity to common fibular nerve (GB-34); one over sinus tarsi and lateral ligaments of ankle mortise (GB-40). Needles will be inserted approximately 1-2cm, connected for 10 min at 2Hz to electrical stimulation (ITO ES-130, 500 ohm test load, 1 to 500Hz). Needles will disposed of in sharps container. Area will be wiped with long handled cotton swab, pressure will be applied for 2 seconds. Subjects will be asked to slowly get up from table and return to lab for second balance assessment.
  Other Names: Electroacupuncture
  Arms: Electroacupuncture
Device: Streitberger placebo needles (Asia-Med, 0.03 x 30 mm) — As with experimental group, controls will do balance assessment pre- and post-intervention. Streitberger placebo needles (Asia-Med, 0.03 x 30 mm), blunted with a telescoping mechanism, will be used. Subjects will feel slight prick, and shaft will telescope into handle, creating illusion of skin penetration. Needles will be held in place by plastic ring covered by a bandage. They are validated for blinding. They will be placed over non-traditional acupuncture points on medial aspect of leg, in direct opposition to treatment group needles. Needle placement is not intended to produce therapeutic outcome. The needles will be connected to a wire, which will be turned on for 10 minutes but no stimulation will be felt.
  Arms: Control

SUMMARY:
Introduction: Ankle sprains, the most common sports-related musculoskeletal injury, account for approximately 25% of sports injuries. An estimated 40% of these individuals will progress to develop chronic functional ankle instability (CFAI), which can significantly affect athletic performance and activities of daily life. Stresses from the injury can damage the ligaments, muscles, nerves and mechanoreceptors. It is widely accepted that ankle proprioception is critical for balance and that individuals with CFAI demonstrate decreased proprioception and altered muscular function, which impairs postural stability. The goal of this study is to determine if a single application of electroacupuncture can have an immediate positive outcome related to balance in individuals with CFAI.

Methods: This single blinded randomized trial will include 12 subjects receiving a single application of electroacupuncture and 12 subjects in the placebo group receiving sham electroacupuncture. Subjects aged 18-50 with a history of unilateral inversion ankle sprain(s) and chronic symptoms of instability will be selected. Balance will be assessed pre- and post-treatment using force plate data during a single-leg stance and via the Star Excursion Balance Test (SEBT). GB-34 and GB-40 will be used for the experimental group and non-traditional points on the medial aspect of the leg will be used for the sham electroacupuncture group. Both will be connected to the electrical stimulation unit for 10 minutes. Results from this study may inform future research investigating the ability of EA at decreasing the risk of ankle sprains, improving perceived stability, and reducing the risk of subsequent degenerative changes.

DETAILED DESCRIPTION:
A single application of electroacupuncture improves balance greater than placebo control in subjects with chronic functional ankle instability

Specific Aim #1:

Evaluate the effect of a single application of electroacupuncture on center of pressure mean total velocity in individuals with chronic functional ankle instability during single-leg stance compared to placebo control.

H0: EA will not improve postural sway during single-leg stance compared to placebo control.

Specific Aim #2:

Describe the effects of a single application of EA compared to placebo on mean total displacement, as well as the mediolateral and anterioposterior components during single-leg stance for possible trends to inform hypothesis generation.

Specific Aim #3:

Correlate the results from the Star Excursion Balance Test with results of the single-leg stance measures to inform hypothesis generation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* History of inversion ankle sprains
* Chronic symptoms of instability

Exclusion Criteria:

* Please see inclusion criteria

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Tests of single-leg standing | 10 seconds
  Tests of single-leg standing balance have been demonstrated to have moderate to excellent group reliability, and therefore are being utilized to compare the balance performance of subjects with chronic functional ankle instability

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Rowan, DC, Principal Investigator — Canadian Memorial Chiropractic College
Locations (1):
- Canadian Memorial Chiropractic College, Toronto, Ontario, Canada